CLINICAL TRIAL: NCT02370875
Title: Combined Effects of rTMS and Botulinum Toxin in Benign Essential Blepharospasm: A Novel Approach
Brief Title: rTMS and Botulinum Toxin in Benign Essential Blepharospasm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201400993
Record Dates: First submitted 2015-02-10; First posted 2015-02-25 (Estimated); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Benign Essential Blepharospasm
MeSH Terms: conditions — Benign essential blepharospasm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Real rTMS stimulation (Experimental): Repetitious transcranial magnetic stimulation (rTMS) will be delivered using the Magstim RapidStim2 over each anterior cingulate cortex, using a figure-of-eight coil. The investigators will apply rTMS with 0.2 Hz frequency to the ACC. 180 stimuli will be delivered with a stimulator output of 100% active motor threshold (AMT). AMT will be assessed at the tibialis anterior muscle with the coil. The AMT will be defined as the lowest stimulation intensity required to evoke a 150 μV potential in the target muscle. To determine the stimulation site for ACC, the coil will be placed over Fz and then moved over the midline of the brain in 0.5-cm steps anteriorly, until the point of maximum motor evoked potential in the orbicularis oculi (OO) muscle. The coil position will be marked on the skin. These rTMS sessions will be repeated daily for 10 days.
  Interventions: Device: Magstim RapidStim2
- Sham rTMS Stimulation (Sham Comparator): During sham repetitious transcranial magnetic stimulation (rTMS), subjects will undergo the same procedure for identifying stimulus location as used in patients receiving real rTMS using the sham Magstim RapidStim2 coil. This coil will be placed on the patient's head in an identical manner however will not be connected to the Magstim device. Instead another coil will be connected to provide stimulation sound. In each stimulation condition, the Magstim will be placed behind the patient and not visible to him or her. Placebo sham coil which produces discharge noise and vibration similar to a real coil without stimulating the cerebral cortex. During rTMS, all patients will continue to wear ear plugs as instructed during the real stimulation sessions.
  Interventions: Device: Sham Magstim RapidStim2

INTERVENTIONS:
Device: Magstim RapidStim2 — Application of repetitious transcranial magnetic stimulation (TMS) pulses using Magstim RapidStim2 to a specific brain target at predefined stimulation parameters.
  Arms: Real rTMS stimulation
Device: Sham Magstim RapidStim2 — Same procedure as real rTMS without stimulating the cerebral cortex.
  Arms: Sham rTMS Stimulation

SUMMARY:
Benign essential blepharospasm (BEB) is a functionally disabling focal dystonia. Botulinum neurotoxin (BoNT) therapy is suboptimal in many BEB patients. Repetitious transcranial magnetic stimulation (rTMS) therapy is a promising noninvasive therapy and has shown positive benefits in BEB. rTMS therapy can be easily combined with BoNT injections to enhance the effects of BoNT in BEB.

DETAILED DESCRIPTION:
A two week course of rTMS therapy to achieve sustained benefits will be employed. With standard BoNT treatment, the peak-dose benefits are seen at about 4-6 weeks after the administration of injections. rTMS will be introduced during this peak-dose period (about 6 weeks after BoNT or T1).The effects of combined therapy at about 10 weeks after BoNT injections (T2) and at about 12 weeks after BoNT injections (T3) will be examined along with the physiological effects at these time points.

ELIGIBILITY:
Inclusion Criteria:

* subjects diagnosed with blepharospasm or cranio-cervical dystonia who receive BoNT therapy at the Center for Movement Disorders will be approached. The investigators will enroll only those subjects who report experiencing positive benefits with BoNT but lasting about 10 weeks or less.

Exclusion Criteria:

* pregnancy
* active seizure disorder
* significant cognitive impairment
* exposure to neuroleptics
* presence of a metallic body such as pacemaker, implants, prosthesis, artificial limb or joint, shunt, metal rods and hearing aid.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Wagle-Shukla, MD, Principal Investigator — University of Florida
Locations (1):
- Center for Movement Disorders and Neurorestoration, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: sets of eyes
Period: Overall Study
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Started | 6; 6 sets of eyes | 6; 6 sets of eyes
Completed | 6; 6 sets of eyes | 6; 6 sets of eyes
Not Completed | 0; 0 sets of eyes | 0; 0 sets of eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: sets of eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation | Total
Number analyzed (Participants) | 6 | 6 | 12
Number analyzed (sets of eyes) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.8 (7.4) | 69.3 (7.2) | 69.1 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
BEB severity on Jankovic Rating Scale [Mean (Standard Deviation); unit: Score on evaluation] — The Jankovic Rating Scale (JRS) subscore for severity of Essential Blepharospasm. Rated on a 5-point scale (0-4) where a higher score equals higher severity of BEB.
  Score on evaluation | 3.1 (0.1) | 2.5 (1.1) | 2.8 (0.5)
BEB frequency on Jankovic Rating Scale [Mean (Standard Deviation); unit: Score on evaluation] — The Jankovic Rating Scale (JRS) subscore for frequency of Essential Blepharospasm. Rated on a 5-point scale (0-4) where a higher score equals higher frequency of blinking due to BEB.
  Score on evaluation | 3.3 (0.7) | 2.6 (1.2) | 2.9 (0.8)
BEB blink frequency on video rating [Mean (Standard Deviation); unit: Blinks per minute] — An eye blink is defined as any visible, bilateral, and synchronous contraction of the orbicularis oculi (OO muscle), causing eyelid drop. Blink frequency will be expressed as blinks per minute and will be determined from a 5 minute video.
  Blinks per minute | 38.7 (15.2) | 37 (16.7) | 37.9 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in JRS Severity Score
Description: The change in the score of the Jankovic Rating Scale subscore for severity. Rated on a 5-point scale (0-4), where a higher score indicates higher severity of blepharospasm.
Time Frame: 2 weeks after rTMS
Measure: Mean (Standard Deviation); unit: Change in score
Units Other Than Participants: sets of eyes
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Number analyzed (Participants) | 6 | 6
Number analyzed (sets of eyes) | 6 | 6
Change in score | -1.8 (0.8) | -0.1 (0.23)

2. Primary Outcome: Change in JRS Frequency Score
Description: The change in the score of the Jankovic Rating Scale subscore for frequency. Rated on a 5-point scale (0-4), where a higher score indicates higher frequency of forced blinks in blepharospasm.
Time Frame: 2 weeks after rTMS
Measure: Mean (Standard Deviation); unit: Change in score
Units Other Than Participants: sets of eyes
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Number analyzed (Participants) | 6 | 6
Number analyzed (sets of eyes) | 6 | 6
Change in score | -1.4 (0.8) | -0.1 (0.2)

3. Primary Outcome: Change in Number of Sustained Forced Eye Blinks
Description: A video recording (5 minutes) was scored by two blinded neurologists to count the number of sustained forced eye-blinks.
Time Frame: 2 weeks after rTMS
Measure: Mean (Standard Deviation); unit: blinks per 5 minutes
Units Other Than Participants: sets of eyes
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Number analyzed (Participants) | 6 | 6
Number analyzed (sets of eyes) | 6 | 6
blinks per 5 minutes | -2.3 (0.8) | -0.5 (0.1)

4. Primary Outcome: Change in Duration of Forced Blinks
Description: A video recording (5 minutes) was scored by two blinded neurologists to count the duration of sustained forced eye-blinks.
Time Frame: 2 weeks after rTMS
Measure: Mean (Standard Deviation); unit: Change in seconds
Units Other Than Participants: sets of eyes
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Number analyzed (Participants) | 6 | 6
Number analyzed (sets of eyes) | 6 | 6
Change in seconds | -2.6 (1.1) | -0.3 (0.8)

5. Secondary Outcome: Change in CDQ-24 QOL Score
Description: Change in score of the Craniocervical dystonia questionnaire (CDQ-24), a self-reported questionnaire designed to evaluate the impact of dystonia on activities of daily living and quality of life. The total CDQ-24 score can therefore range from 0 to 96, with higher scores meaning greater impairment due to dystonia.
Time Frame: 2 weeks after rTMS
Population: Score from self-reported questionnaire
Measure: Mean (Standard Deviation); unit: Change in score
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Number analyzed (Participants) | 6 | 6
Change in score | -10.6 (5.1) | -4.3 (2.1)

6. Secondary Outcome: Change in CDQ-24 ADL Subscore
Description: Change in Actitivities of Daily Living (ADL) subscore of the Craniocervical dystonia questionnaire (CDQ-24), a questionnaire designed to evaluate quality of life outcomes for patients with dystonia. The ADL subscore is obtained from 6 of the 24 questions. Each question is rated on a 5-point scale (0-4), where a higher number indicates increasing severity of impairment for that daily activity due to dystonia. The total ADL subscore takes the sum of the number from five questions (a value from 0 to 24), then linearly transforms that sum to a 0-100 scale, where a higher score means greater impairment in daily life.
Time Frame: 2 weeks after rTMS
Measure: Mean (Standard Deviation); unit: Change in score
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Number analyzed (Participants) | 6 | 6
Change in score | -30 (12.1) | -15 (13.2)

7. Secondary Outcome: Change in Social Subscale of CDQ-24
Description: Change in the social subscore of the Craniocervical dystonia questionnaire (CDQ-24), a questionnaire designed to evaluate quality of life outcomes for patients with dystonia. The social subscore is obtained from 4 of the 24 questions. Each question is rated on a 5-point scale (0-4), where a higher number indicates increasing severity of social impairment due to dystonia. The total social subscore can therefore range from 0 to 16, with higher scores meaning greater impairment of social activities.
Time Frame: 2 weeks after rTMS
Measure: Mean (Standard Deviation); unit: Change in score
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Number analyzed (Participants) | 6 | 6
Change in score | -15 (11.2) | -2.5 (13.2)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT02370875/Prot_SAP_000.pdf